CLINICAL TRIAL: NCT03366701
Title: Association Between Automatic Psychological Processes, Self-regulatory Capacities and Physical Activity and Sedentary Behaviors Adoption, Change and Maintenance Among Persons With Chronic Diseases
Brief Title: Motivational Parameters Associated With Physical Activity and Sedentary Behaviors Among Persons With Chronic Diseases
Status: Completed | Type: Observational
Sponsor: 5 Santé (Other)
Responsible Party: Sponsor
Other Study IDs: 5S_AUTAP
Record Dates: First submitted 2015-12-30; First posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Health Behavior
Keywords: physical activity; sedentary behavior; implicit attitudes; self regulation; intention; chronic diseases
MeSH Terms: conditions — Health Behavior; Motor Activity; Sedentary Behavior; Self-Control; Chronic Disease | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patient during rehabilitation program: Patient performing a 5 weeks inpatient pulmonary rehabilitation program
  Interventions: Other: Rehabilitation
- Patient after the rehabilitation program: Patient in their domicile after the 5 weeks program
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — The intervention (routine care) correspond to five weeks rehabilitation program

SUMMARY:
The principal aim of these researches is to explored the role of motivational parameters, including: automatic and controlled psychological processes and self-regulatory capacities, in physical activity and sedentary behaviors adoption and maintenance. Precisely investigators are interested in change in motivational and self-regulatory processes during rehabilitation programs and their prospective influences on self-reported and objective behaviors among persons with chronic diseases.

DETAILED DESCRIPTION:
Automatic processes refered to implicit attitudes measured through the implicit association test (IAT) and single category (SC-IAT). Controlled processes refered to the variables of the Theory of Planned Behavior measured by questionnaire. Self regulatory capacities refered to the concept of impulsivity measured by questionnaire and executive functions measured through the STROOP task and Wisconsin Card Sorting Task.

Physical activity and sedentary behaviors are measured by questionnaire and accelerometry.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Under health care coverage

Exclusion Criteria:

* medical contra-indication to exercise
* concerned by acute health procedure
* enable to completed computerised tests and questionnaires
* Under psychiatric treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Person with chronic illness such cardio-respiratory and metabollic diseases
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Objective physical activity and sedentary behaviors | This measure will be performed 6 months after the program during one week.
  Objective physical activity and sedentary behaviors are measured with accelerometers. Time spent in sedentary behaviors (less than 1,5 Metabolic equivalents) ; light physical activity (1,5 to 3 Mets), moderate physical activities (3 to 6 Mets) and high intensities (up to 6 Mets) are recorded by the monitors.

SECONDARY OUTCOMES:
automatic psychological processes associated to physical activity and sedentary behaviors | At the inclusion (T0)
  Automatic processes : implicit association test (IAT, Greenwald et al., 1998). Reaction time and percentage of errors is using for the scoring procedure. The score is comprised between -2 and +2.
controlled psychological processes associated to physical activity and sedentary behaviors | At the inclusion (T0)
  Controlled processes: variables of the Theory of Planned Behavior measured by questionnaire (Likert scale 1 to 7 point). 4 scores comprise between 1 to 7.
Executive functions | At the inclusion (T0) and 6 months after
  Executive functions: the STROOP task and Wisconsin Card Sorting Task (WCST) design on computer. For the STROOP task a subtraction of the mean reaction time of two specifics blocks is computed (unity: millisecond). The WCST provide a score in percentage of errors.
Self-regulatory capacities | at the inclusion (T0)
  Self-regulatory capacities: impulsivity measured by questionnaire, a score comprise between 20 (low score of impulsivity) and 80 is computed.
Self-report sedentary behavior | this measure will be performed 6 months after the program
  Self-report Sedentary Behavior is measured by questionnaire. The score reflect a cumulative score in hour / week..
Self-report physical activity | this measure will be performed 6 months after the program
  Self-report physical activity is measured by questionnaire. The scoring procedure requires to make the sum of the frequency by week (0 to 7days/weeks) with a score in minutes for those activities (1 point : less to 15 min ; 2 point : 16 to 30 ; 3 point : 31 to 60 ; 4 point : more than 60).

CONTACTS AND LOCATIONS:
Overall Officials: Nelly HERAUD, Ph-D, Study Director — 5 Santé
Locations (1):
- Chevance, Montpellier, Herault, France